CLINICAL TRIAL: NCT05777421
Title: Efficacy of Virtual Reality Based Exercise Regimes on Kinesiophobia, Pain and Functional Disability in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/5
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthristis
Keywords: Range of Motion, Proprioception

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy along with Natural apophyseal glides and the second will receive Natural Apophyseal Glides in addition to cranial base release with conventional physical therapy. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy Regime for Knee Osteoarthrithis (Active Comparator): Pt will receive conventional therapy targeting stretching and stretching of knee musculature in combination with electrotherapy for pain modulation.
  Frequency : 2-3 times for a duration of 6 weeks Pt will be guided home plan based exercises.
  Interventions: Procedure: Conventional Physical Therapy for Knee Osteoarthriths
- Virtual reality Based Therapeutic Exercise Regimes (Experimental): VR-based therapeutic exercise regimes utilizing Xbox, that focus on different activities like Partial squatting, lunges, side lunge, calf raises, and hamstring curls.
  Gaming exercises begin will an easy warm up round and get challenging with different rounds of each game as the patient progresses to week 6.
  Frequency: 2-3 times for a duration for 6 weeks Pt will be guided home plan based exercises
  Interventions: Procedure: Virtual Reality-Based Therapeutic Exercise regimes

INTERVENTIONS:
Procedure: Conventional Physical Therapy for Knee Osteoarthriths — Participants of Group A will receive the conventional physical therapy for Knee Osteoarthistis for a duration of 6 weeks atleast 2 times a week
  Arms: Conventional Physical Therapy Regime for Knee Osteoarthrithis
Procedure: Virtual Reality-Based Therapeutic Exercise regimes — * Participants of Group B will receive Virtual Reality Based therapeutic exercises on the Xbox. The difficulty level of the games will progess each week. The duration of training will also also progress at treatment week progresses.
  * Frequency: 2-3 times a week for 6 weeks. Minimum 12 sessions in total.
  Arms: Virtual reality Based Therapeutic Exercise Regimes

SUMMARY:
Knee Osteoarthritis is one of the most prevalent degenerative conditions in Pakistan. Although a variety of Physical therapy treatments have been proven to be beneficial in patients with early stages of knee Osteoarthritis. However, a few secondary impairments like Kinesiophobia which is the fear of movement have been unaddressed. Usually after conventional physical therapy, patients find immediate or short-term relief and that leads to cessation of follow up sessions. In situations like these, kinesiophobia is the greatest threat to mobility and can eventually effect quality of life by decreasing functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral knee OA involving mediolateral compartment
* Knee OA grade 2
* Aged 40-65 years
* Both Male and Female
* NPRS value greater than

Exclusion Criteria:

* Patients with history of
* History of systemic disorder (e.g., rheumatoid arthritis, ankylosing spondylitis).
* History of malignancy.
* History of trauma.
* Previous knee surgery.
* Congenital musculoskeletal deformity (e.g., scoliosis, kyphosis).
* Patients with history of fracture
* Patients with history of Chondropatella Malacia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 6 weeks
  Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia
Pain intensity | 6 weeks
  Will be Measured using the Numeric Pain rating scale
Functional Disability | 6 weeks
  Will be measured using WOMAC Osteoarthritis Index

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan